CLINICAL TRIAL: NCT07237958
Title: Effects on the Olfactory Epithelium in the Nose and the Olfactory Nerve (Nervus Olfactorius) From Exposure to Diesel Exhaust
Brief Title: Effects on the Olfactory Epithelium and the Olfactory Nerve From Exposure to Diesel Exhaust
Acronym: DINOSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umeå University (Other)
Collaborators: University Hospital, Umeå (Other); University of Eastern Finland (Other); Czech Academy of Sciences (Other)
Responsible Party: Principal Investigator, Ala Muala, MD, PhD, Umeå University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: 2018-438-31; x (Other Grant/Funding Number: The Swedish Research Council)
Record Dates: First submitted 2025-07-04; First posted 2025-11-20 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Alzheimer Disease (AD); Dementia Alzheimer Type; Air Pollution Exposure
Keywords: cognitive function; Alzheimer Disease; Diesel Exhaust; Olfactory nerve
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exposure to diesel exhaust (Active Comparator): The participants will be exposed in an exposure chamber for diesel exhaust in a concentration of 300 µg/m³ for one hour.
  Interventions: Other: Diesel Exhaust Particles
- Exposure to filtered air (Placebo Comparator): The participants will be exposed in an exposure chamber to filtered air for one hour.
  Interventions: Other: Filtered air

INTERVENTIONS:
Other: Diesel Exhaust Particles — During exposure to diesel exhaust, participants alternate between 15-minute periods of rest and exercise on an ergometer cycle with a workload that results in a minute ventilation of 20L/min/m² body surface area. Symptom recording is done every 30 minutes, following a routine based on a modified Borg scale.
  Arms: Exposure to diesel exhaust
Other: Filtered air — During exposure to filtered air, participants alternate between 15-minute periods of rest and exercise on an ergometer cycle with a workload that results in a minute ventilation of 20L/min/m² body surface area. Symptom recording is done every 30 minutes, following a routine based on a modified Borg scale
  Arms: Exposure to filtered air

SUMMARY:
The goal of this study is to study the effect exposure to air pollution and its effect on development of dementia.

Does the diesel exhaust change the function of the olfactory system?

Have the exposures measurable effects on the sense of smell and cognitive ability?

Forty people are exposed to diesel exhaust exhaust and filtered air. The exposures are blinded and in a randomized order. Both groups undergo biopsies of the olfactory epithelium in the nose under local anesthesia after the exposures and after performing cognitive test.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* non-smoker

Exclusion Criteria:

* Allergic rhinitis
* Asthma
* Diabetes mellitus
* Kidney or liver failure
* Angina pectoris or previous ventricular arrhythmia
* Systolic blood pressure >190 mmHg or <100 mmHg
* Previous blood disease
* Blood donation in the last three months prior to study start
* Previous or ongoing tobacco smoking and exposure to air pollution in the workplace
* Absence of informed consent

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2023-05-12 (Actual); Study Completion 2023-05-19 (Actual)

PRIMARY OUTCOMES:
Diesel exhaust causes cellular dysfunction of the olfactory system | 3 years.
  RNA sequencing and DNA methylation will be conducted to identify biomarkers for acute exposure to diesel exhaust.

SECONDARY OUTCOMES:
Cognitive test | 3 years
  Olfactory function well be evaluated by using "sniffin' sticks," and a Letter-Digit Substitution Test as a marker for cognitive processing speed.

CONTACTS AND LOCATIONS:
Locations (1):
- Umeå Univeristy, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Martikainen MV, Aakko-Saksa P, van den Broek L, Cassee FR, Carare RO, Chew S, Dinnyes A, Giugno R, Kanninen KM, Malm T, Muala A, Nedergaard M, Oudin A, Oyola P, Pfeiffer TV, Ronkko T, Saarikoski S, Sandstrom T, Schins RPF, Topinka J, Yang M, Zeng X, Westerink RHS, Jalava PI. TUBE Project: Transport-Derived Ultrafines and the Brain Effects. Int J Environ Res Public Health. 2021 Dec 28;19(1):311. doi: 10.3390/ijerph19010311. PMID 35010571
- See also: ADAIR website — https://www.alzheimer-europe.org/our-work/past-work/past-projects/adair?language_content_entity=en

DOCUMENTS (2):
  • Study Protocol (2021-06-17): https://cdn.clinicaltrials.gov/large-docs/58/NCT07237958/Prot_000.pdf
  • Informed Consent Form (2021-06-17): https://cdn.clinicaltrials.gov/large-docs/58/NCT07237958/ICF_001.pdf